CLINICAL TRIAL: NCT00329758
Title: Phase II Study of Rosuvastatin´s Effect on Amnesia and Orientation Through Galveston Outcome Amnesia Test in Humans With Moderate Head Injury
Brief Title: Effect of Rosuvastatin on Amnesia and Orientation Through Galveston Outcome Amnesia Test in Moderate Head Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other); AstraZeneca (Industry)
Responsible Party: Humberto Tapia
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26-06ROHI
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2009-03

CONDITIONS: Head Injury
Keywords: moderate head injury; rosuvastatin; statin; amnesia; orientation
MeSH Terms: conditions — Craniocerebral Trauma; Amnesia; Orientation, Spatial | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: rosuvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rosuvastatin — 20 mg oral, during 10 days
  Other Names: Crestor
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether rosuvastatin is effective in the management of moderate head injury by improving amnesia and orientation.

DETAILED DESCRIPTION:
The head injury is a frequent problem of health, which produces high morbid-mortality. Today is the main cause of death and disability between 18 and 40 years. In addition it originates expensive expenses in health care systems.

Head injury produces damage by primary mechanisms related to impact, then by biochemical ways which are activated and they carry to secondary damage. Many studies have been conducted for explaining secondary injury, the majority conclude there is a kind of ischemic lesion related maybe with changes in cerebral flow and metabolism. The management today is trying to avoid progression in secondary damage without good outcome. Many drugs and measures has been ineffective.

In the last years has been demonstrated in head injury microvascular damage like stroke. Statins o inhibitors of HMG CoA reductase are drugs used in dyslipidemia, frequently for reduction in LDL. Experimental and clinical studies in stroke have shown improvement in outcome. The toxicity related to statin is myopathy and hepatopathy, both with low incidence without fatal cases. Rosuvastatin has been postulated be the most powerful with longest life and toxicity similar to another statins.

We have designed this study for demonstrate if the administration of rosuvastatin in the first 24 hours and by 10 days has improvement in amnesia and orientation, furthermore outcome.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman >16 and <50 years with HI less 24 hours in progression and Glasgow between 9 y 12.
* Man or woman >16 and <50 years with HI and Glasgow l3, with lesions in TC scan.
* Acceptance of family to participate (first grade).

Exclusion Criteria:

* History of HI with disability
* History of neurological or psychiatric disease with disability.
* Administration 24 hrs previous of: fibrates, niacin, ciclosporin, azoles, macrolides, inhibitors of protease, nefazodone, verapamil, diltiazem,amiodarone.
* Existence of systemic injury with life in compromise (massive bleeding, exposition of bone in fracture, hepatic or splenic laceration or in great vessels and shock).
* Administration of THAM, mannitol, barbiturates, corticosteroids, scavengers of free radicals, inhibitors of lipidic peroxidation, indometacin, calcium antagonist, antagonists of neurotransmitters
* Existence of intracranial lesion which needs surgery.
* Lesions not classifiable or in brainstem.
* Allergy to the drug.
* Hepatopathy or myopathy (or) history of this, or clinical data of hepatic disease.
* Management previous in other Hospital.
* Pregnancy

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Galveston Orientation and Amnesia Test | Days in be positive

SECONDARY OUTCOMES:
Functional outcome by Disability Rating Scale | at 0 (release) and 3 months
Cytosines (Il-1B, IL-6, TNF-alfa) | Basal and day 3
acute renal Insuficience | Periode of medication (10 days)
Lesion on CT scan | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Torres-Corzo, Neurosurgeon, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"; Humberto Tapia-Perez, MD, Principal Investigator — Facultad de Medicina UASLP
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Tapia-Perez H, Sanchez-Aguilar M, Torres-Corzo J, Rodriguez-Leyva I, Herrera-Gonzalez LB. [Statins and brain protection mechanisms]. Rev Neurol. 2007 Sep 16-30;45(6):359-64. Spanish. PMID 17899518
- [Background] Tapia-Perez J, Sanchez-Aguilar M, Torres-Corzo JG, Gordillo-Moscoso A, Martinez-Perez P, Madeville P, de la Cruz-Mendoza E, Chalita-Williams J. Effect of rosuvastatin on amnesia and disorientation after traumatic brain injury (NCT003229758). J Neurotrauma. 2008 Aug;25(8):1011-7. doi: 10.1089/neu.2008.0554. PMID 18690806
- [Background] Tapia-Perez JH, Sanchez-Aguilar M, Schneider T. The role of statins in neurosurgery. Neurosurg Rev. 2010 Jul;33(3):259-70; discussion 270. doi: 10.1007/s10143-010-0259-4. Epub 2010 Apr 29. PMID 20429022